CLINICAL TRIAL: NCT01353599
Title: Acute and Chronic Effects of Inhaled Steroids on Pulmonary Function in Persons With Spinal Cord Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, Miroslav Radulovic, M.D., Staff Physician, VA Office of Research and Development
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01349
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Tetraplegia; Pulmonary Function
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asmanex (Experimental): Study participants will receive inhaled Mometasone Furoate (Asmanex) 220mcg once daily for 8 weeks.
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Mometasone furoate — 220mcg once daily, for eight weeks
  Other Names: Asmanex

SUMMARY:
Individuals with chronic cervical SCI are known to have a restrictive ventilatory defect due to complete or partial loss of respiratory muscle innervation which is dependent upon the level and completeness of injury [2]. In addition, they share many aspects of obstructive airway physiology commonly associated with asthma. In asthma, physiological responses such as decrease in baseline airway caliber, bronchodilatation following inhalation of a beta-2-adrenergic agonist or anticholinergic agent, airway hyperreactivity, are all closely related to airway inflammation. The cause of such inflammation is unclear, and may be multi-factorial and attributable to: recurrent respiratory infections due to inability to effectively clear secretions, unopposed parasymphathetic innervation, and loss of functional sympathetic innervation to the airways. Therefore, the investigators propose to test for the possible involvement the above mechanisms by pharmacological intervention, and to study effects of such intervention on overall pulmonary function and indirect measures of pulmonary inflammation: levels of FeNO, exhaled breath condensate (EBC) inflammatory biomarker profile, pulmonary function tests, and cellular profile of the induced sputum.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old; and
* Stable, tetraplegia C3-C8 levels (duration of injury >1 year).

Exclusion Criteria:

* Smoking, active or history of smoking during the last six months
* Active respiratory disease(s), such as COPD, inflammatory lung disease, obstructive lung diseases, or acute respiratory infections
* No known history of asthma during lifetime or recent (within 3 months) respiratory infections;
* Ventilator dependence;
* Use of medications known to affect the respiratory system, such as nizoral;
* aldesleukin
* oral corticosteroids (e.g., prednisone, dexamethasone)
* natalizumab
* drugs affecting liver enzymes that remove mometasone from your body (such as azole antifungals including itraconazole, macrolide antibiotics including erythromycin, cimetidine, rifamycins including rifabutin, St. John's wort, certain anti-seizure medicines including carbamazepine)
* Use of medications known to alter airway caliber;
* Coronary heart and/or artery disease, as indicated in the patient medical record;
* Hypertension, baseline blood pressure ≥ 140/90mHg;
* Adrenal insufficiency, as indicated in the patient medical record;
* Pregnancy;
* Lack of mental capacity to give informed consent;
* History of glaucoma;
* History of cataracts; and
* Persisting pressure ulcer, or a recently healed wound (e.g., ≤3 months since wound closure).
* History of a milk protein allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The Acute and Chronic Effects of an Inhaled Corticosteroid on Pulmonary Function | 1 Hour
  The following measures of pulmonary function will be assessed (At baseline and eight weeks post intervention):
  Spirometry Body Plethysmography

SECONDARY OUTCOMES:
The Effects of an Inhaled Corticosteroid on Biomarkers of Inflammation in Exhaled Breath Condensate | 30 mins, baseline and 8 week post
  Biomarkers of inflammation will be assessed from measured exhaled breath condensates collected at baseline and 8 weeks post.
The Effect of an Inhaled Corticosteroid on the cellular profile of induced sputum | 15 mins during, baseline and 8 week post
  We will determine the effects of the inhaled corticosteroid on the cellular profile of sputum. Sputum will be collected and centrifuged, then viewed under a microscope for determination of cellular profile.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Radulovic, MD, Principal Investigator — James J. Peters VA Medical Center
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York